CLINICAL TRIAL: NCT05289453
Title: Phacoemulsification in Acute Congestive Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hany Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Hany Mahmoud, principal investigator, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-22-02-29
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): patients wit acute congestive glaucoma and treated bt lens extraction by phacoemulsification after IOP control
  Interventions: Procedure: lens extraction by phacoemulsification

INTERVENTIONS:
Procedure: lens extraction by phacoemulsification — lens extraction by phacoemulsification

SUMMARY:
Acute primary angle closure (APAC) is usually caused by an abrupt closure of the trabecular meshwork in the anterior chamber angle that leads to a sudden rise in intraocular pressure (IOP). APAC is a subgroup of angle closure disease characterised by a sudden onset of headache, blurred vision, seeing halos around lights, corneal oedema, mid-dilated pupil, eye pain and redness. Asian also has a much higher incident rate of APAC compare to the Caucasian population - with the crude incidence rate of 12.2 and 10.4 per 100,000 people per year in the above 30-year-old population of Singapore and Hong Kong, respectively . This is higher than the average incidence rate of 3.9-4.1 cases per 100,000 people per year in the European regions .

In APAC, both LPI and primary lens extraction by phacoemulsification and intraocular lens implant (phaco/IOL) were demonstrated to be effective to control IOP elevation. The latter has been shown to be the more effective treatment than LPI for IOP reduction at the early and mid-term IOP control. Together with the advancement of phaco/IOL technique, primary lens extraction is the more popular choice of treatment nowadays. However, operating on an eye with early aborted APAC is technically challenging and may increase the risk of complications because of the presence of corneal oedema, inflammation, shallow anterior chamber, floppy iris and unstable lens. Furthermore, "the best time window" for performing lens extraction after an APAC attack remains uncertain. The long-term results (e.g. more than 5 years) of early lens extraction compared to the conventional LPI are also unknown. In this study, we summarise the approach of treating APAC at the initial acute stage and review the studies that consider IOP control in the mid and long term. We would also touch on the role of goniosynechialysis, trabeculectomy and endoscopic cyclophotocoagulation in treating APAC, as well as considering the economic aspect of treatment.

Aim of the study: to evaluate the safety and efficacy of phacoemulsificatiojn in cases of acute congestive glaucoma

ELIGIBILITY:
Inclusion Criteria:

* patients with acute congestive glaucoma

Exclusion Criteria:

* people under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
iop control | 3 months follow-up
  iop will be assessed by applination tonometry and the values will be recorded, the success is defined by normal iop values during follow up period (3 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Hany Mahmoud, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after research completion